CLINICAL TRIAL: NCT03276507
Title: Multisystem Shortness of Breath Evaluation Study
Acronym: MUSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, LUIS SEIJO MACEIRAS, Attending Physician, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Other Study IDs: EO 113/2016_FJD
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea | interventions — Echocardiography; Electrocardiography; Diagnostic Imaging; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Pulmonary function studies
Diagnostic Test: Echocardiogram
Diagnostic Test: Electrocardiogram
Diagnostic Test: Chest radiography
Diagnostic Test: Blood test
Behavioral: Quality of life questionnaire

SUMMARY:
The MUSE study is a prospective observational cohort study of patients referred to pulmonary and/or cardiology specialty clinic for evaluation of shortness of breath or dyspnea. Patients will undergo all pertinent testing and will be required to fill out a number of epidemiologic and quality of life related questionnaires. Follow up will continue for at least one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to Pulmonary and/or Cardiology clinic for the evaluation of unexplained dyspnea.

Exclusion Criteria:

* Patients with a known cause of dyspnea such as established cardiopulmonary disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing evaluation for dyspnea in a specialized clinic (Pulmonary and/or Cardiology)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Dyspnea etiology | 3 months
  All patients will undergo cardiopulmonary testing and will be offered quiestionnaires including the M3 online questionnaire

SECONDARY OUTCOMES:
Quality of Life | 6 months
  Several questionnaires will be used including the M3 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: German Peces-Barba, MD, Principal Investigator — Fundación Jimenez Díaz
Locations (1):
- Fundación Jimenez Díaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No